CLINICAL TRIAL: NCT07178977
Title: Psychoeducation for Parents of Adolescents With Anorexia Nervosa as a Supportive Treatment Approach
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PPO-ZD-MH
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Eating Disorders; Anorexia Nervosa
Keywords: eating disorders; Anorexia Nervosa; Parental Stress; Parental Coping
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Masking Description: The nature of the intervention (Psychoeducation and waitlist groups) makes it impossible to mask interventions assigned.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Psychoeducation for parents of adolescents with anorexia nervosa (Experimental): Parents in the intervention group will participate in a structured four-week psychoeducation program designed to support families of adolescents with anorexia nervosa. The program consists of four weekly group sessions, each lasting 90 minutes, delivered at the Child Psychiatry Department, University Medical Centre Ljubljana. Each session follows a standardized format: (1) review of homework and discussion of experiences, (2) introduction of the session content, (3) structured psychoeducational module, and (4) assignment of new tasks.
  Interventions: Behavioral: Psychoeducation group
- Waitlist control group (Active Comparator): Parents in the waitlist control group will continue with treatment as usual and will not participate in the psychoeducation program during the first month of the study. They will complete baseline and one-month assessments while waiting. After this one-month period, the waitlist group will receive the same structured four-week psychoeducation program as the intervention group.
  Interventions: Behavioral: Psychoeducation group

INTERVENTIONS:
Behavioral: Psychoeducation group — A structured, group-based psychoeducation program designed for parents of adolescents with anorexia nervosa. The intervention consists of four weekly sessions, each lasting 90 minutes, delivered in small groups (up to 7 families) at the Child Psychiatry Department, University Medical Centre Ljubljana. Each session follows a standardized structure. The session topics are: Understanding eating disorders; Maintaining factors in anorexia nervosa and strategies to address them; Establishing and supporting normal eating patterns, Promoting and sustaining change.
  The program is adapted from evidence-based approaches, including family-based treatment (FBT) and enhanced cognitive-behavioral therapy (CBT-E), and is tailored to a psychoeducational group format for parents. The aim is to reduce parental distress, improve coping, and enhance adolescent treatment outcomes (BMI, eating disorder symptoms, anxiety, depression).

SUMMARY:
This randomized controlled trial will evaluate the effectiveness of a structured four-week psychoeducation program for parents of adolescents diagnosed with anorexia nervosa (AN). The program aims to improve parental coping and improve adolescent treatment outcomes.

Seventy adolescents with AN (ages 11-19) and their parents will be recruited at the University Medical Centre Ljubljana, Slovenia. Families will be randomly assigned to either an intervention group, receiving immediate psychoeducation, or a waitlist control group, receiving the program after one month. The psychoeducation program consists of four weekly 90-minute sessions covering eating disorder characteristics, maintaining factors, strategies for normal eating, and approaches for supporting change.

Primary outcomes include change in adolescent body mass index (BMI) from baseline to post-intervention and three-month follow-up. Secondary outcomes include adolescent symptoms of eating disorders, anxiety, and depression, as well as parental anxiety, depression, stress, social support, and self-efficacy. The study will test whether early, structured parental involvement through psychoeducation improves both adolescent clinical outcomes and parental coping.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a severe psychiatric disorder with high morbidity and mortality, typically emerging during adolescence. Effective treatment requires family involvement, yet parents frequently experience high levels of stress, anxiety, guilt, and isolation while supporting their child through treatment. Psychoeducation for parents may reduce parental distress and simultaneously enhance adolescent treatment outcomes, but rigorous randomized trials are limited.

This randomized controlled trial will evaluate a structured four-week psychoeducation program for parents of adolescents diagnosed with anorexia nervosa (AN). The intervention is designed to complement treatment as usual and is based on principles from enhanced cognitive-behavioral therapy for eating disorders (CBT-E) and existing psychoeducational protocols. The program aims to improve parental coping skills, reduce parental psychological distress, and improve adolescent treatment outcomes.

Families will be recruited from the Child Psychiatry Department at the University Medical Centre Ljubljana, Slovenia. After providing informed consent, families will be randomized into either:

Intervention group - parents receive immediate participation in the psychoeducation program while their adolescents continue treatment as usual, or

Waitlist control group - parents continue treatment as usual and receive the program after one month.

Each psychoeducation group will include parents of up to seven adolescents and will meet weekly for four sessions, each lasting 90 minutes. Session structure includes: review of previous homework, introduction of new material, core psychoeducational content, and assignment of new tasks. Topics progress from understanding eating disorder characteristics and myths, to identifying maintaining factors, establishing normal eating patterns, and promoting sustainable behavioral and emotional change.

Both adolescents and parents will complete assessments at defined time points. Adolescents will be evaluated for changes in body mass index (BMI) and self-reported psychological symptoms, while parents will be assessed for anxiety, depression, stress, perceived social support, and self-efficacy. The intervention group will be assessed at baseline, immediately post-intervention, and three months after the program, while the waitlist control group will complete assessments at baseline and one month later, prior to receiving the intervention.

The primary outcome is change in adolescent BMI from baseline to post-intervention. Secondary outcomes include changes in adolescent eating disorder symptoms, anxiety, and depression, as well as parental psychological well-being and coping. The study will use a waitlist-controlled design to isolate the effects of the psychoeducation program and will monitor whether improvements are sustained at three-month follow-up.

The trial is expected to provide evidence on the role of structured parental psychoeducation as an adjunct to standard treatment for adolescent AN and to offer a scalable model for integrating family-focused interventions into child and adolescent mental health services.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 11-19 years
* Clinical diagnosis of anorexia nervosa (AN) according to DSM-5 criteria
* Referred for treatment at the Child Psychiatry Department, Pediatric Clinic, University Medical Centre Ljubljana
* At least one parent/legal guardian willing to participate in the psychoeducation program
* Signed informed consent by parent(s) and assent from adolescent

Exclusion Criteria:

* Adolescents with severe comorbid psychiatric conditions requiring alternative treatment (e.g., psychosis, severe intellectual disability, active substance dependence)
* Adolescents or parents unable to understand Slovenian language sufficiently to participate in group sessions or complete questionnaires
* Families already engaged in a structured psychoeducation or similar parent-support program at the time of recruitment

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Adolescent Body Mass Index (BMI) | Baseline (T1), Post-intervention (4 weeks, T2), Follow-up (3 months post-intervention, T3).
  Body weight and height will be measured and BMI will be calculated (kg/m²). Change in BMI will be assessed as an indicator of treatment response.

SECONDARY OUTCOMES:
Change in Eating Disorder Symptoms - Eating Disorder Examination Questionnaire (EDE-Q 6.0) | Baseline (T1), Post-intervention (4 weeks, T2), Follow-up (3 months post-intervention, T3).
  Self-reported eating disorder symptoms will be assessed using the Eating Disorder Examination Questionnaire, Version 6.0 (EDE-Q 6.0). The questionnaire includes four subscales: Restraint, Eating Concern, Shape Concern, and Weight Concern, and produces a global score. Each item is rated on a 7-point scale (0-6), where higher scores indicate more severe eating disorder symptoms. The global score is the average of all items, with 0 representing no symptoms and 6 representing the most severe level of symptoms.
Change in Anxiety and Depression Symptoms - Revised Child Anxiety and Depression Scale (RCADS - Youth Version) | Baseline (T1), Post-intervention (4 weeks, T2), Follow-up (3 months post-intervention, T3).
  Self-reported symptoms of anxiety and depression will be assessed using the Revised Child Anxiety and Depression Scale (RCADS). The questionnaire consists of 47 items, each rated on a 4-point scale (0-3), where 0 = never, 1 = sometimes, 2 = often, and 3 = always. Higher scores indicate greater severity of anxiety or depression symptoms.
  The RCADS includes six subscales: Separation Anxiety, Social Phobia, Generalized Anxiety Disorder, Panic Disorder, Obsessive-Compulsive Disorder, and Depression, as well as total anxiety and total internalizing scores.
Change in Parental Anxiety and Depression - Hospital Anxiety and Depression Scale (HADS) | Baseline (T1), Post-intervention (4 weeks, T2), Follow-up (3 months post-intervention, T3).
  Self-reported symptoms of anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS). The questionnaire consists of 14 items, with 7 items assessing anxiety and 7 items assessing depression. Each item is rated on a 4-point scale (0-3), where 0 represents no symptoms and 3 represents the most severe level of symptoms. Higher scores indicate greater severity of anxiety or depression.
  Each subscale (Anxiety and Depression) has a total score range of 0-21, with higher scores reflecting worse psychological distress.
Change in Parental Stress - Perceived Stress Scale (PSS-10) | Baseline (T1), Post-intervention (4 weeks, T2), Follow-up (3 months post-intervention, T3).
  Perceived stress will be assessed using the 10-item Perceived Stress Scale (PSS-10). The questionnaire consists of 10 items, each rated on a 5-point scale (0-4), where 0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, and 4 = very often. Higher scores indicate greater perceived stress.
  The total score ranges from 0 to 40, with 0 representing no perceived stress and 40 representing the highest level of perceived stress.
Change in Parental Self-Efficacy - General Self-Efficacy Scale (GSE) | Baseline (T1), Post-intervention (4 weeks, T2), Follow-up (3 months post-intervention, T3).
  General self-efficacy will be assessed using the General Self-Efficacy Scale (GSE). The questionnaire consists of 10 items, each rated on a 4-point scale (1-4), where 1 = not at all true, 2 = hardly true, 3 = moderately true, and 4 = exactly true.
  The total score ranges from 10 to 40, with higher scores indicating greater perceived self-efficacy, reflecting a better outcome.
Change in Parental Perceived Social Support - Multidimensional Scale of Perceived Social Support (MSPSS). | Baseline (T1), Post-intervention (4 weeks, T2), Follow-up (3 months post-intervention, T3).
  Perceived social support will be assessed using the Multidimensional Scale of Perceived Social Support (MSPSS). The questionnaire consists of 12 items, each rated on a 7-point scale (1-7), where 1 = very strongly disagree and 7 = very strongly agree.
  The total score ranges from 12 to 84, with higher scores indicating greater perceived social support, which reflects a better outcome. The MSPSS also provides subscale scores for support from family, friends, and significant others.
Parent-Reported Adolescent Anxiety and Depression - Revised Child Anxiety and Depression Scale - Parent Version (RCADS-P) | Baseline (T1), Post-intervention (4 weeks, T2), Follow-up (3 months post-intervention, T3).
  Parent-reported symptoms of adolescent anxiety and depression will be assessed using the Revised Child Anxiety and Depression Scale - Parent Version (RCADS-P). The questionnaire consists of 47 items, each rated on a 4-point scale (0-3), where 0 = never, 1 = sometimes, 2 = often, and 3 = always. Higher scores indicate greater severity of adolescent anxiety or depression symptoms as perceived by parents.
  The RCADS-P provides six subscale scores: Separation Anxiety, Social Phobia, Generalized Anxiety Disorder, Panic Disorder, Obsessive-Compulsive Disorder, and Depression, as well as total anxiety and total internalizing scores.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Kodrič, PhD, Study Director — Unit of Child Psychiatry, University Children's hospital, University Medical Centre Ljubljana; Marija Anderluh, PhD, Study Chair — Unit of Child Psychiatry, University Children's hospital, University Medical Centre Ljubljana
Locations (1):
- Unit of Child Psychiatry, University Children's hospital, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
It is planned to publish it on the repository of University of Ljubljana. Personal data will not be provided, participants will be encrypted and unrecognizable.
Supporting Information: Study Protocol
Time Frame: After the study will be finished

REFERENCES:
- [Background] Winn S, Perkins S, Murray J, Murphy R, Schmidt U. A qualitative study of the experience of caring for a person with bulimia nervosa. Part 2: Carers' needs and experiences of services and other support. Int J Eat Disord. 2004 Nov;36(3):269-79. doi: 10.1002/eat.20068. PMID 15478136
- [Background] Macdonald P, Murray J, Goddard E, Treasure J. Carer's experience and perceived effects of a skills based training programme for families of people with eating disorders: a qualitative study. Eur Eat Disord Rev. 2011 Nov-Dec;19(6):475-86. doi: 10.1002/erv.1065. Epub 2010 Dec 28. PMID 22021124
- [Background] Lee H, Desai S, Choi YN. Improvements in Quality of Life and Readiness for Change After Participating in an Eating Disorder Psychoeducation Group: A Pilot Study. Int J Group Psychother. 2024 Jul;74(3):268-303. doi: 10.1080/00207284.2024.2341293. Epub 2024 May 10. PMID 38727719
- [Background] Konstantellou A, Sternheim L, Hale L, Simic M, Eisler I. The experience of intolerance of uncertainty for parents of young people with a restrictive eating disorder. Eat Weight Disord. 2022 May;27(4):1339-1348. doi: 10.1007/s40519-021-01256-8. Epub 2021 Jul 22. PMID 34292530
- [Background] Hudson JI, Hiripi E, Pope HG Jr, Kessler RC. The prevalence and correlates of eating disorders in the National Comorbidity Survey Replication. Biol Psychiatry. 2007 Feb 1;61(3):348-58. doi: 10.1016/j.biopsych.2006.03.040. Epub 2006 Jul 3. PMID 16815322
- [Background] Honey A, Boughtwood D, Clarke S, Halse C, Kohn M, Madden S. Support for parents of children with anorexia: what parents want. Eat Disord. 2008 Jan-Feb;16(1):40-51. doi: 10.1080/10640260701773447. PMID 18175232
- [Background] Hillege S, Beale B, McMaster R. Impact of eating disorders on family life: individual parents' stories. J Clin Nurs. 2006 Aug;15(8):1016-22. doi: 10.1111/j.1365-2702.2006.01367.x. PMID 16879546
- [Background] Hibbs R, Rhind C, Leppanen J, Treasure J. Interventions for caregivers of someone with an eating disorder: a meta-analysis. Int J Eat Disord. 2015 May;48(4):349-61. doi: 10.1002/eat.22298. Epub 2014 May 31. PMID 24891101
- [Background] Fursland A, Erceg-Hurn DM, Byrne SM, McEvoy PM. A single session assessment and psychoeducational intervention for eating disorders: Impact on treatment waitlists and eating disorder symptoms. Int J Eat Disord. 2018 Dec;51(12):1373-1377. doi: 10.1002/eat.22983. PMID 30584661
- [Background] Fletcher L, Trip H, Lawson R, Wilson N, Jordan J. Life is different now - impacts of eating disorders on Carers in New Zealand: a qualitative study. J Eat Disord. 2021 Jul 23;9(1):91. doi: 10.1186/s40337-021-00447-z. PMID 34301344
- [Background] Dalle Grave R, Eckhardt S, Calugi S, Le Grange D. A conceptual comparison of family-based treatment and enhanced cognitive behavior therapy in the treatment of adolescents with eating disorders. J Eat Disord. 2019 Dec 31;7:42. doi: 10.1186/s40337-019-0275-x. eCollection 2019. PMID 31893120
- [Background] Coelho JS, Suen J, Marshall S, Burns A, Lam PY, Geller J. Parental experiences with their child's eating disorder treatment journey. J Eat Disord. 2021 Jul 27;9(1):92. doi: 10.1186/s40337-021-00449-x. PMID 34315529
- [Background] Carpita B, Muti D, Cremone IM, Fagiolini A, Dell'Osso L. Eating disorders and autism spectrum: links and risks. CNS Spectr. 2022 Jun;27(3):272-280. doi: 10.1017/S1092852920002011. Epub 2020 Nov 9. PMID 33161925
- [Background] Bezance J, Holliday J. Mothers' experiences of home treatment for adolescents with anorexia nervosa: an interpretative phenomenological analysis. Eat Disord. 2014;22(5):386-404. doi: 10.1080/10640266.2014.925760. Epub 2014 Jul 14. PMID 25024015
- [Background] Agras WS. The consequences and costs of the eating disorders. Psychiatr Clin North Am. 2001 Jun;24(2):371-9. doi: 10.1016/s0193-953x(05)70232-x. PMID 11416936